CLINICAL TRIAL: NCT05922787
Title: The Effect of Reiki on Sexual Function and Sexual Self-Confidence in Women With Sexual Distress
Brief Title: The Effect of Reiki on Sexual Function and Sexual Self-Confidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sümeyye Barut, Assit. Prof, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/3795
Record Dates: First submitted 2023-06-16; First posted 2023-06-28 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Therapeutic Touch; Sexuality
Keywords: reiki; sexual distress; sexual self-confidence; sexual experience
MeSH Terms: conditions — Sexuality | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial
Who Masked: Participant
Masking Description: This study was designed as a randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Personal Information Form, Female Sexual Distress Scale-Revised (FSD-R),Arizona Sexual Experiences Scale (ASEX),Sexual Self-Confidences Scale (SSS) were utilized for the collection of research data. First of all, FSD-R was applied to the women, and the women who obtained a score above11.5 points or more from the FSD-R were invited to the study.Then, the Personal Information Form, ASEX, and SSS were first applied to the women invited to the study. Women in the experimental group received Reiki once a week for four weeks. No initiative was applied to the pregnant women in the control group. The FSD-R, ASEX and SSS were applied to all participant women after four weeks following the first application. The application of the measurement tools took 10-15 minutes.
  Interventions: Other: Reiki
- Control (No Intervention): The researchers applied no initiative to the control group, and the women in the control group solely had the routine checks. The women in the control group filled out all pretest forms(Personal Information Form, FSD-R, ASEX, SSS. The post-test forms (FSD-R, ASEX, SSS) were re-administered 4 weeks later to women who did not receive any intervention.

INTERVENTIONS:
Other: Reiki — In the study, women received four Reiki sessions once a week for four weeks from the researchers with Usuı Shiki Ryoho Reiki 1
  Arms: Experimental

SUMMARY:
Background and Purpose: This study aimed to determine the effect of Reiki on sexual function and sexual self-confidence in women with sexual distress.

Materials and Methods: This randomized controlled study was conducted with women between the ages of 15-49 years who were registered at a family health center in the eastern region of Turkey and had sexual distress. The sample of the study consisted of 106 women, 53 in the experimental group and 53 in the control group. Women in the experimental group received Reiki once a week for four weeks, while no intervention was applied to those in the control group. Data were collected using the Female Sexual Distress Scale-Revised (FSDS-R), the Arizona Sexual Experiences Scale (ASEX), and the Sexual Self-confidence Scale (SSS).

DETAILED DESCRIPTION:
2. Methods 2.1. Research Design and Sample In this randomized controlled study, participants were randomly assigned to the experimental (Reiki group) or control groups. The study was conducted using women between the ages of 15-49 years who were registered at a Family Health Center in a province of eastern Turkey. This primary healthcare center provides reproductive health services to women such as family planning, education, and counseling, and includes 3 family physicians and 3 family health workers (midwives and/or nurses). The center was randomly selected considering its socioeconomic environment, proximity to the city center, and registered number of women. The center serves approximately 21,000 people, including around 1600 women. Additionally, there is a quiet and peaceful room in the center to hold Reiki sessions. Women who agreed to participate in the study and met the study inclusion criteria were included in the study.

The study inclusion criteria were as follows: being a woman, scoring 11.5 or above on the Female Sexual Distress Scale-Revised (FSDS-R), and being sexually active during the study. The study exclusion criteria were as follows: being pregnant or postpartum, having a diagnosis of any psychiatric illness or sexual dysfunction.

The sample size was determined using OpenEpi (Open Source Epidemiologic Statistics for Public Health) version 3.1, a web-based program. A priori power analysis was performed to estimate the appropriate sample size. As the primary outcome of the study, the mean sexual life score was determined to be 13.70 (with a standard deviation of 5.48) in the literature review. The sample size was calculated as 53 for each group (53 for the experimental group and 53 for the control group) assuming a 5% two-tailed type I error rate, 95% confidence interval, 80% power to represent the population, and a 3-point increase in sexual life score after the intervention.

To reach the sample size, a total of 200 women were evaluated for eligibility criteria. Of them, 47 did not meet the inclusion criteria and 25 refused to participate in the study. In addition, 13 out of 67 women in the experimental group were excluded from the study as they did not continue to participate in Reiki sessions, while 8 out of 61 women in the control group were excluded from the study because they did not want to continue participating in the study. The study was completed with a total of 106 women, 53 in the experimental group and 53 in the control group.

2.2. Randomization Women who agreed to participate in the study and met the inclusion criteria were randomly assigned to experimental and control groups in the order of their arrival at the Family Health Center. A randomization was performed using the Random Integer Generator method, which can be found in the Numbers subsection of the random.org website. Single-column tables were created using numbers from 1 to 106 (https://www.random.org/). Women who referred to the Family Health Center were randomly assigned to numbers 1 and 2 in the column, considering the numbers 1 and 2. The decision of which number would correspond to the experimental or control group was determined by drawing lots. The number 1 was assigned to the experimental group and the number 2 to the control group.

2.3. Data Collection Tools 2.3.1. Personal Information Form The form was created by the researchers and includes questions about women's some introductory characteristics (age, education level, family type, income level, and employment status).

2.3.2. Female Sexual Distress Scale-Revised (FSDS-R) The FSDS-R assesses various aspects of sexual distress in women, including subjective stress and psychological impact associated with sexual dysfunction and is used to identify women with and without sexual dysfunction. The scale consists of 13 items on a five-point Likert scale ranging from never (0) to always. Total scale score ranges between 0 and 52. A higher score indicates higher levels of sexual distress. A cutoff score of ≥11.5 has been recommended to detect the presence of sexually-related personal distress in Turkish women. The Cronbach's alpha reliability coefficient of the scale was found as 0.86 by Aydın et al., while it was determined as 0.78 in this study.

2.3.3. Arizona Sexual Experiences Scale (ASEX) The ASEX assess changes and disorders in sexual function. It was validated in Turkish in 2004. This six-point Likert type scale consists of five items on sexual desire, psychological arousal, physiological arousal (vaginal lubrication), orgasmic capacity, and orgasmic pleasure. Each item is scored from 1 to 6, with a total score ranging from 5 to 30. A lower score indicates a stronger, easier, and more satisfying sexual response, while a higher score suggests sexual dysfunction. The Cronbach's alpha reliability coefficient of the scale was found as 0.89, while it was determined as 0.73 in this study.

2.3.4. Sexual Self-confidences Scale (SSS) The SSS was developed in Turkish by Çelik and validated for its reliability and validity. This four-point Likert type scale consists of 13 items to measure sexual self-confidence. Each item is scored from never (1) to always. Total scale score ranges between 13 and 52. A higher score indicates higher levels of sexual self-confidence. The Cronbach's alpha reliability coefficient of the scale was found as 0.88, while it was determined as 0.78 in this study.

2.4. Data Collection In the study, pre-test data were collected from women through face-to-face interviews in the counseling room at the FHC using a questionnaire that included introductory information as well as the scales used in the study. The same method was used to collect post-test data after four weeks of the intervention. The scales lasted around 10-15 minutes to complete.

2.5. Intervention In the study, women received four Reiki sessions once a week for four weeks from the researchers with Usuı Shiki Ryoho Reiki 1 (Degree 1). The researchers received training and certification in Reiki techniques before starting the intervention. In Reiki 1, the practitioner provides healing through touch or by holding hands a few centimeters above the body, establishing "aura harmony" between the practitioner and the person receiving the treatment. No studies have established what the "energy" referred to in Reiki is; a belief in Reiki is an unsubstantiated belief, rather than an established fact. Reiki practitioners use Reiki with light-hand contact to facilitate an opening of their patients' and their own "energy channels.". Reiki practitioners have explained that the body has seven chakras (at the head, between the eyes, the throat, the chest, the abdominal cavity, the groin, and the upper hip). The sessions were conducted individually in the counseling rooms of the FHC. Each session lasted for 30-40 minutes. The most important rule in Reiki practice for participants is to allow the practitioner to facilitate the flow of energy. It is not necessary for the person receiving Reiki to believe in it because Reiki is universal life energy and is present in everyone. The following sequence is generally applied in Reiki protocols: 1. Before beginning Reiki, the practitioner and the patient remove any jewelry on their bodies. 2. The patient can sit on a chair or lie down on a treatment table with arms and legs open on both sides of the body. 3. It is not necessary to remove the patient's clothes, and their body can be covered with a sheet or a blanket. 4. Reiki is applied by placing hands on the patient's body or holding them a few centimeters above their body. 5. The practitioner sends energy to each chakra or area on the body for 3-5 minutes, depending on the flow of energy, and this time can extend up to 10-20 minutes.6. The practitioner washes their hands. 7. The process is recorded. In addition to the general protocol of Reiki, the practitioner in this study preferred a quiet room and dimmed the lights to prevent distractions. Each woman started the practice lying on her back, fully dressed, with her eyes closed, arms and legs straight and palms facing upwards. At the beginning of the Reiki practice, the practitioner held her hands 2-3 centimeters above each woman's body and made circular movements from her head to her feet to adjust her aura. After this "aura alignment" process, the practitioner placed her hands directly on each woman's body. The practice was performed from top to bottom, starting from the head and spending 3-5 minutes in each hand position at each of the seven main chakras. Each position was held for between one to five minutes, or until the Reiki practitioner felt the energy stop flowing. However, since Reiki application can be done for a longer period on the area where discomfort is felt, and also since the area of sexuality is located in the root chakra, the application of Reiki was ended with a total of 30-40 minutes, with an extra 10 minutes on the root chakra.

No intervention was applied to women in the control group by the researcher; and they only received the service they needed from the FHC.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman,
* Scoring 11.5 or above on the Female Sexual Distress Scale-Revised (FSDS-R)
* Being sexually active during the study.

Exclusion Criteria:

* being pregnant or postpartum
* having a diagnosis of any psychiatric illness or sexual dysfunction

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women between the ages of 15-49 years
Enrollment: 106 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Female Sexual Distress Scale-Revised (FSDS-R) | Change from Sexual Distress at 4 weeks
  The FSDS-R was assesses various aspects of sexual distress in women, including subjective stress and psychological impact associated with sexual dysfunction and is used to identify women with and without sexual dysfunction. The scale consists of 13 items on a five-point Likert scale ranging from never (0) to always. Total scale score ranges between 0 and 52. A higher score indicates higher levels of sexual distress. A cutoff score of ≥11.5 has been recommended to detect the presence of sexually-related personal distress in Turkish women.

SECONDARY OUTCOMES:
Arizona Sexual Experiences Scale (ASEX) | Change from Sexual Experiences at 4 weeks
  The ASEX assess changes and disorders in sexual function. It was validated in Turkish in 2004. This six-point Likert type scale consists of five items on sexual desire, psychological arousal, physiological arousal (vaginal lubrication), orgasmic capacity, and orgasmic pleasure. Each item is scored from 1 to 6, with a total score ranging from 5 to 30. A lower score indicates a stronger, easier, and more satisfying sexual response, while a higher score suggests sexual dysfunction.
Sexual Self-confidences Scale (SSS) | Change from Sexual Self-confidences at 4 weeks
  This four-point Likert type scale consists of 13 items to measure sexual self-confidence. Each item is scored from never (1) to always. Total scale score ranges between 13 and 52. A higher score indicates higher levels of sexual self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat University, Elâzığ, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No